CLINICAL TRIAL: NCT03765580
Title: The Influence of Fish Consumption on Polyunsaturated Fatty Acid (PUFA) Status (iFish Study)
Brief Title: The Influence of Fish Consumption on Polyunsaturated Fatty Acid (PUFA) Status
Acronym: iFish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: University of Rochester (Other); Lund University (Other); Ministry of Health, Republic of Seychelles (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REC/16/0077
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Polyunsaturated Fatty Acid (PUFA) Status
Keywords: Polyunsaturated fatty acids (PUFA); fish; fish consumption; women; childbearing age
MeSH Terms: interventions — In Situ Hybridization, Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): No fish
  Interventions: Other: Control
- 1 portion of fish per week (Experimental): 140g fish/week
  Interventions: Dietary Supplement: Fish
- 2 portions of fish per week (Experimental): 280g fish/week
  Interventions: Dietary Supplement: Fish

INTERVENTIONS:
Dietary Supplement: Fish — Lunch containing fish
  Arms: 1 portion of fish per week; 2 portions of fish per week
Other: Control — Lunch containing no fish
  Arms: Control group

SUMMARY:
Polyunsaturated fatty acids (PUFA) are important for health, for example for the immune system, heart health and the brain. PUFA are found in fish, nuts and oils; including these foods in the diet provides the body with PUFA. The body can also produce some PUFA in a series of steps. It has been found that genetics influences the levels of PUFA produced in the body. This study will investigate whether fish consumption influences PUFA status in women of childbearing age when accounting for FADS genotype by conducting a controlled human intervention study. Participants will be asked to consume none, one or two portions of oily fish per week for 8 weeks and their response in PUFA status measured. This study will also use collected blood, hair, urine and faecal samples collected from the intervention study to explore other biomarkers of fish consumption. The aim of this study is to investigate whether fish consumption influences PUFA status in women of childbearing age when accounting for FADS genotype and to explore the potential of a novel biomarker, using hair MeHg:δ34S values, to accurately predict fish consumption. The study will initially involve providing a buccal swab sample which will investigate genes which are related to fatty acids. The participant will provide a buccal swab sample so that their genotype can be determined. The researcher who will contact the participant once genotype has been determined to arrange a baseline appointment. Participants will attend the Human Intervention Studies Unit at Ulster University, Coleraine once or twice weekly for a period of 8 weeks where they will receive lunch. This lunch will contain either tuna, sardines, or no fish depending on the intervention group you will be allocated to. Examples of lunch time meals they may receive include sandwiches, baked potato or salad which will include the type of fish they have been allocated to receive. Those allocated to the no fish group will receive a fish free alternative lunch. Participants will be asked to continue to follow their normal diet and lifestyle over the intervention period of 8 weeks. All participants will attend a baseline and post intervention appointment where they will have weight, height and body composition measured. Participants will also complete questionnaires to provide medical, lifestyle and dietary information. All participants will be asked to provide a sample of blood, urine, hair and faeces to assess biomarkers of fish consumption at baseline and post intervention appointments. Collected blood, urine, hair and faecal samples will be analysed for biomarkers of fish consumption. Participants will also be asked to return to the Human Intervention Studies Unit (HISU) 8 weeks after the intervention study has been completed (week 16) to provide a third hair sample and complete a Fish Feedback Questionnaire. In the 8 wks following conclusion of the study they will be free to return to their normal diet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females - premenopausal, child-bearing age, not planning to become pregnant
* Age 18-45years old
* Low consumers of fish (<2 portions/ week) or those willing to reduce their fish consumption one month prior to commencing the study to the equivalent of 2 portions per month or less
* Willing to eat 1 or 2 portions (140 grams or 280 grams) of either tuna or sardines per week for a period of 8 weeks
* Not consuming fish oil supplements
* Not consuming protein supplements
* Not allergic to seafood

Exclusion Criteria:

* Regularly eat fish or not willing to do washout period where they reduce fish consumption
* Are allergic to seafood
* Are taking fish oil supplements or are taking protein supplements
* Are pregnant or menopausal
* Have very short hair (a small section of hair, approximately 200 strands, will be taken at the nap of the neck for analysis purposes)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 49 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Polyunsaturated fatty acid (PUFA) status | Change at 8 weeks from baseline
  Serum Polyunsaturated fatty acid (PUFA) status

SECONDARY OUTCOMES:
Hair mercury | Change at 8 & 16 weeks from baseline
  Hair mercury status
Lipid profile | Change at 8 weeks from baseline
  Serum lipid profile
Iodine | Change at 8 weeks from baseline
  Urine iodine
Inflammatory status | Change at 8 weeks from baseline
  Cytokine concentration (Interleukin (IL)-5, IL-1β, IL-2, IL-4, IL-6, IL-10, MCP-1, TARC, sFlt-1, VEgF-D, CRP, TNF-α, IFN-γ)
Oxidative stress | Change at 8 weeks from baseline
  Change in glutathione peroxidase and 8-isoprostanes
Microbiota | Change at 8 weeks from baseline
  Faecal microbiota profile
Thyroid hormones | Change at 8 weeks from baseline
  Serum T3, T4 and thyroid-stimulating hormone (TSH). Dried blood spot for thyroglobulin, T4 and TSH
Stable isotopes | Change at 8 & 16 weeks from baseline
  Hair methyl-mercury and sulphur-34
Methyl-mercury (MeHg) | Change at 8 weeks from baseline
  Whole blood and urine MeHg

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Co.Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Conway MC, McSorley EM, Mulhern MS, Spence T, Wijngaarden EV, Watson GE, Wahlberg K, Pineda D, Broberg K, Hyland BW, Cobice DF, Strain JJ, Yeates AJ. The influence of fish consumption on serum n-3 polyunsaturated fatty acid (PUFA) concentrations in women of childbearing age: a randomised controlled trial (the iFish Study). Eur J Nutr. 2021 Apr;60(3):1415-1427. doi: 10.1007/s00394-020-02326-w. Epub 2020 Jul 28. PMID 32725293